CLINICAL TRIAL: NCT03838068
Title: Clinical and Radiographic Evaluation of Pulpotomy Technique for Preserving Vitality of Traumatized Anterior Permanent Immature Teeth: A Randomized Clinical Trial
Brief Title: Pulpotomy Technique Preserving Vitality of Traumatized Anterior Permanent Immature Teeth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gihan M Abuelniel ,PhD (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Gihan M Abuelniel ,PhD, Associate Professor of Pediatric Dentistry, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19118
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Pulp Exposure, Dental
Keywords: trauma; vital immature; MTA; Biodentine
MeSH Terms: conditions — Dental Pulp Exposure; Wounds and Injuries | interventions — tricalcium silicate; mineral trioxide aggregate; Pemetrexed; Procaine

STUDY DESIGN:
Intervention Model Description: Access cavity in traumatized central incisors will be assigned into experimental or control group using simple randomization 1:1 by the help of the computer software(random.org).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients and their parents, the assessor and the statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mineral trioxide aggegate (Active Comparator): white mineral trioxide aggregate (MTA) calcium silicate-based cement
  Interventions: Biological: mineral trioxide aggregate; Procedure: cervical pulpotomy; Drug: Local Anesthetics Procaine
- Biodentine (Experimental): calcium silicate-based cement that consists of tricalcium silicate, dicalcium silicate, calcium carbonate, calcium oxide, zirconium oxide, and CH.
  Interventions: Biological: Biodentine; Procedure: cervical pulpotomy; Drug: Local Anesthetics Procaine

INTERVENTIONS:
Biological: Biodentine — Biodentine is considered a calcium silicate cement
  Other Names: Calcium silicate-based
  Arms: Biodentine
Biological: mineral trioxide aggregate — calcium based silicate cement
  Other Names: MTA
  Arms: Mineral trioxide aggegate
Procedure: cervical pulpotomy — coronal pulp tissue was removed till the orifice
Drug: Local Anesthetics Procaine — 40 mg/0.01 mg/ml contains sodium metabisulfite and sodium and articaine as an active substance
  Other Names: artinibsa

SUMMARY:
Aim of the study: To compare the clinical and radiographic outcomes of mineral trioxide aggregate (MTA) and Biodentine as vital pulp therapy materials (pulpotomy) preserving the vitality of traumatized immature anterior permanent teeth.

Materials and Methods: fifty vital traumatized immature anterior permanent teeth exposed with symptomatic /asymptomatic pulpitis were included in the study according to inclusion criteria and were equally divided in two groups. Included teeth were randomly assigned to either a control group (MTA 25 teeth) or a test group (Biodentine 25 teeth). After conducting pulpotomy and covering pulp stumps with the MTA and Biodentine, treated teeth received permanent restorations. Blinded clinical and radiographic evaluations were performed at different time intervals (base line immediate postoperative, 6, 12 and 18 months) according to clinical and radiographic criteria of success. Data were recorded and analyzed.

DETAILED DESCRIPTION:
Informed consent was obtained from all patients prior to treatment, and patients were offered Root canal treatment in case of treatment failure.

Thirty-three patients who were referred to the postgraduate pediatric dentistry department clinic for the management of their traumatized permanent incisors teeth were assessed. Only Patients who had a traumatic incisor tooth with a vital pulp (detected by clinical signs/symptoms) were included.

Incisors were assigned randomly in the two groups. The MTA group was considered the control group while the biodentine was the test group.

All patients who were clinically eligible for enrollment in the study went through screening pre-operative digital periapical radiographic examination to assess the degree of root development/ formation and any dental infections or anomalies that could interfere with the planned treatment.

The main investigator performed all pulpotomies. Local anesthesia was administrated followed by rubber dam isolation, the coronal pulp tissue was excised to the level of the orifice using a diamond bur with water cooling. Hemostasis was achieved by gentle placement of a saline-moistened cotton pellet over amputated pulps for 5-10 min. Pulp stumps were covered with:

In the first group (control group) white mineral trioxide aggregate (MTA) ProRoot® MTA (Dentsply/ Johnson City,TN,USA) was used as the reference material for comparison and was prepared according to the manufacturer's instructions. A 3-mm-thick layer of MTA was placed over the amputated pulps and was gently adapted to the dentinal walls using a wet cotton pellet deep onto the radicular pulp. A self-cure glass ionomer (GC; GC Corporation, Tokyo, Japan) was placed over the pulpotomy agent before final restoration of composite resin (ClearﬁlTM, Kuraray, New York, USA) was done.

In the second group Calcium silicate-based BiodentineTM (Septodont Ltd., Saint Maur des Fausse´s, France) was mixed according to the manufacturer's instructions, pulpotomy was performed, radicular pulp was covered, and teeth received self-cure glass ionomer prior to final restoration with the same technique as in the first group.

ELIGIBILITY:
Inclusion Criteria:

* The patient age range 7.5-9 years.
* Noncontributory medical history
* Unilateral/ and or bilateral central incisors tooth with complicated trauma (exposure size ≥ 1mm)
* The tooth should give positive response to cold testing
* Clinical diagnosis of reversible pulpitis without periapical rarefaction
* The tooth is restorable, mobility was within normal limits
* No signs of pulpal necrosis including sinus tract or swelling

Exclusion Criteria:

* Teeth with mature roots
* Signs and symptoms of irreversible pulpitis
* Non-restorable teeth
* Negative response to cold testing, the presence of sinus tract or swelling
* No pulp exposure
* Bleeding could not be controlled after full pulpotomy in 6 minutes

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
presence of pain,sensitivity to percussion/ palpation | 18 months
  by asking the patient( questionnaire) (Binary measure) ( Yes or No) where Yes indicates failure of the treatment
Swelling or sinus tract | 18 months
  by visual examination (binary measure)( Yes or No) where Yes indicates clinical failure of the treatment
presence of mobility | 18 months
  by the back of the mirror( Binary measure) (Yes or No) where Yes indicates clinical failure of the treatment.

SECONDARY OUTCOMES:
Stage of root development | 18 months
  by radiographic parallel technique ( four root development stages are assessed E, F,G and H) where E is the worse and H is the best stage.
Presence of radiolucency | 18 months
  by radiographic parallel technique (Binary measure) (Yes or No) where Yes indicates radiographic failure of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gihan M Abuelniel, Principal Investigator — Cairo University
Locations (1):
- Gihan Abuelniel, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT03838068/Prot_SAP_000.pdf